CLINICAL TRIAL: NCT03378206
Title: Comparison of the Outcomes of the Treatment of Semiepiphysiodesis Using Hinged and Conventional 8-figure Plates: A Randomized Controlled Clinical Trial
Brief Title: Hinged Versus Conventional 8 Plate for Correction of Genu Valgum or Varum
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Ziming Zhang, Deputy director of Department of Pediatric Orthopedics, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XH-17-013
Record Dates: First submitted 2017-09-25; First posted 2017-12-19 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Genu Valgum or Varum; Growth; Arrested, Bone; Epiphyseal Arrest, Lower Leg
Keywords: genu valgum or varum; eight-plate; epiphysis arrest; hemiepiphysiodesis
MeSH Terms: conditions — Genu Valgum; Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hinged 8-figure plate (Experimental): Hinged 8-figure plate is a novel devise that has modifications in order to improve the treatment effect of conventional 8-figure plate. This arm will be used to verify the effectiveness and feasibility of the modification.
  Interventions: Device: hinged 8-figure plate
- conventional 8-figure plate (Active Comparator): Conventional 8-figure plate is widespread method to treat genu varum and valgus. This arm, as a comparator, will be the control group to verify the feasibility of the novel hinged 8-figure plate.
  Interventions: Device: conventional 8-figure plate

INTERVENTIONS:
Device: hinged 8-figure plate — Hinged 8-figure plate has two arms and a built-in hinge. The rotation of the two arms ranged from 155° to 170° to better fit the contour of the physis in all stages of angular correction. That automatic change can also disperse repeated stress on the surface of periosteum and perichondrium during walking.
  Arms: Hinged 8-figure plate
Device: conventional 8-figure plate — Conventional 8-figure plate is a widespread device to treat angular deformity of lower limbs with moderate successful rate. The device was designed based on the principle of tension band model. It consists of a plate and two screws (epiphyseal screw and metaphyseal screw).
  Arms: conventional 8-figure plate

SUMMARY:
To assess the therapeutic effect of hinged 8-figure plate by comparing with the traditional 8-figure plate through a randomized controlled clinical trial by assessing the differences between preoperative and postoperative data.

The hypothesis is that the hinged 8 plate provides low complications that this treatment is as good as the traditional one.

DETAILED DESCRIPTION:
Angular deformities of the lower limb is major clinical problems encountered in pediatric orthopedics. Deformities can be either valgus or varus and most commonly affect the knee joint, which may result in patella dislocation, gait instability and serious impact on the appearance and function of the lower limbs. Biomechanical studies and gait analysis found that genu varus increased medial articular surface pressure of the knee, while genu valgus increased lateral articular surface pressure, and both of them are the risk factors for osteoarthritis. Surgical treatment techniques include osteotomy and hemiepipysidesis. Osteotomy surgery is the gold standard for severe angular deformity or epiphyseal closed patients, but it was associated with lots of complications, including osteofascial compartment syndrome, neurovascular injury, deep soft tissue infection, nonunion and requiring a long recovery time. While, for patients whose epiphyseal is not closed, the traditional 8 plate hemiepipysidesis has fewer complications. However, it showed some problems in clinical applications, such as steel plate or screw broken. The investigators designed a new hinged 8 plate, which has two arms and a built-in hinge. Based on the previous studies, investigators designed the rotation of the two arms ranged from 155° to 170° to better fit the contour of the physis in all stages of angular correction. That automatic change can also disperse repeated stress on the surface of periosteum and perichondrium during walking. The plate had been tested on animal models that the use of the hinged plate and screw system may be a more reliable technique with minimal complications for correction of angular deformities of the lower limb.

ELIGIBILITY:
Inclusion Criteria:

1. Idiopathic genu valgus or varum
2. Without any treatment
3. lower limb mechanical axis over the tibial plateau in the range of 1/2;
4. Epiphyseal not yet closed, with more than 12 months of growth potential

Exclusion Criteria:

1. Physiological genu valgus or varum
2. Epiphyseal have closed or no growth potential
3. Pathological limb deformity(Blount disease, inflammation,trauma)
4. Other causes of lower limb angular deformity.
5. With surgical contraindications

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2019-09-01 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
The complications. | 2 years
  Surgery related complications including osteofascial compartment syndrome, neurovascular injury, deep soft tissue infection and so on will be observed until correction of deformity.

SECONDARY OUTCOMES:
The corrective rates of medial slope angle. | 2 years
  The angle of medial slope will be measured when reexamination until the correction of deformity, which was used to calculate the corrective rates.
The corrective of Mechanical lateral distal femoral angle. | 2 years
  The corrective of Mechanical lateral distal femoral angle will be measured when reexamination until the correction of deformity. And investigators will calculating the change of this angle.
The movement of two arms of the hinged plate. | 2 years
  The movement of two arms during the experiment will be noted by the changing of two arms angle when reexamination until the correction of deformity.
The residual stress on the implants. | 2 years
  Residual stress (remaining stress of the sample after implant removal) at the rim of the metaphyseal screw hole will be measured using X-ray diffraction.

CONTACTS AND LOCATIONS:
Overall Officials: Ziming Zhang, PhD, Principal Investigator — Department of Pediatric Orthopedics, Xinhua Hospital affiliated to Shanghai Jiao Tong University, School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] BLOUNT WP, CLARKE GR. Control of bone growth by epiphyseal stapling; a preliminary report. J Bone Joint Surg Am. 1949 Jul;31A(3):464-78. No abstract available. PMID 18153890
- [Result] Sharma L, Song J, Felson DT, Cahue S, Shamiyeh E, Dunlop DD. The role of knee alignment in disease progression and functional decline in knee osteoarthritis. JAMA. 2001 Jul 11;286(2):188-95. doi: 10.1001/jama.286.2.188. PMID 11448282
- [Result] Bylski-Austrow DI, Wall EJ, Rupert MP, Roy DR, Crawford AH. Growth plate forces in the adolescent human knee: a radiographic and mechanical study of epiphyseal staples. J Pediatr Orthop. 2001 Nov-Dec;21(6):817-23. PMID 11675562
- [Result] Gottliebsen M, Rahbek O, Poulsen HD, Moller-Madsen B. Similar growth plate morphology in stapling and tension band plating hemiepiphysiodesis: a porcine experimental histomorphometric study. J Orthop Res. 2013 Apr;31(4):574-9. doi: 10.1002/jor.22276. Epub 2012 Nov 28. PMID 23192490
- [Result] Gros DF, Milanak ME, Brady KT, Back SE. Frequency and severity of comorbid mood and anxiety disorders in prescription opioid dependence. Am J Addict. 2013 May-Jun;22(3):261-5. doi: 10.1111/j.1521-0391.2012.12008.x. PMID 23617869
- [Result] Zuege RC, Kempken TG, Blount WP. Epiphyseal stapling for angular deformity at the knee. J Bone Joint Surg Am. 1979 Apr;61(3):320-9. PMID 429399
- [Result] Burghardt RD, Kanellopoulos AD, Herzenberg JE. A technical note on improved instrumentation for Blount staple insertion. J Child Orthop. 2012 Aug;6(4):347-50. doi: 10.1007/s11832-012-0422-2. Epub 2012 Aug 9. PMID 23904903
- [Result] Stevens PM. Guided growth for angular correction: a preliminary series using a tension band plate. J Pediatr Orthop. 2007 Apr-May;27(3):253-9. doi: 10.1097/BPO.0b013e31803433a1. PMID 17414005
- [Result] Burghardt RD, Herzenberg JE, Standard SC, Paley D. Temporary hemiepiphyseal arrest using a screw and plate device to treat knee and ankle deformities in children: a preliminary report. J Child Orthop. 2008 Jun;2(3):187-97. doi: 10.1007/s11832-008-0096-y. Epub 2008 Mar 26. PMID 19308576
- [Result] Boero S, Michelis MB, Riganti S. Use of the eight-Plate for angular correction of knee deformities due to idiopathic and pathologic physis: initiating treatment according to etiology. J Child Orthop. 2011 Jun;5(3):209-16. doi: 10.1007/s11832-011-0344-4. Epub 2011 May 12. PMID 22654982
- [Result] Guzman H, Yaszay B, Scott VP, Bastrom TP, Mubarak SJ. Early experience with medial femoral tension band plating in idiopathic genu valgum. J Child Orthop. 2011 Feb;5(1):11-7. doi: 10.1007/s11832-010-0310-6. Epub 2010 Dec 8. PMID 21415941
- [Result] Driscoll MD, Linton J, Sullivan E, Scott A. Medial malleolar screw versus tension-band plate hemiepiphysiodesis for ankle valgus in the skeletally immature. J Pediatr Orthop. 2014 Jun;34(4):441-6. doi: 10.1097/BPO.0000000000000116. PMID 24172668
- [Result] Aslani H, Panjavy B, Bashy RH, Tabrizi A, Nazari B. The efficacy and complications of 2-hole 3.5 mm reconstruction plates and 4 mm noncanulated cancellous screws for temporary hemiepiphysiodesis around the knee. J Pediatr Orthop. 2014 Jun;34(4):462-6. doi: 10.1097/BPO.0000000000000115. PMID 24172669
- [Result] Lin TY, Kao HK, Li WC, Yang WE, Chang CH. Guided growth by a stainless-steel tubular plate. J Pediatr Orthop B. 2013 Jul;22(4):306-10. doi: 10.1097/BPB.0b013e32835bc42d. PMID 23211739
- [Result] Lee HJ, Oh CW, Song KS, Kyung HS, Min WK, Park BC. Guided growth with a noncannulated screw-plate system for angular deformity of the knee: a preliminary report. J Pediatr Orthop B. 2012 Jul;21(4):339-47. doi: 10.1097/BPB.0b013e3283547198. PMID 22568964
- [Result] Schroerlucke S, Bertrand S, Clapp J, Bundy J, Gregg FO. Failure of Orthofix eight-Plate for the treatment of Blount disease. J Pediatr Orthop. 2009 Jan-Feb;29(1):57-60. doi: 10.1097/BPO.0b013e3181919b54. PMID 19098648
- [Result] Burghardt RD, Specht SC, Herzenberg JE. Mechanical failures of eight-plateguided growth system for temporary hemiepiphysiodesis. J Pediatr Orthop. 2010 Sep;30(6):594-7. doi: 10.1097/BPO.0b013e3181e4f591. PMID 20733426
- [Result] Wu Z, Zhao D, Zhao L, Liu J, Li H, Zhu J, Ma F, Porter DE. A comparison between a hinged plate and screw system and a conventional tension-band plate and screw system used for correction of an angular deformity of the lower limb: an animal study. J Orthop Surg Res. 2015 May 3;10:57. doi: 10.1186/s13018-015-0198-4. PMID 25935152